CLINICAL TRIAL: NCT00944619
Title: Randomised, Two-Period Crossover Study to Assess the Efficacy of Overnight Computer-based Glucose Control Compared With Conventional Pump Therapy Following the Consumption of Alcohol in Adults With Type 1 Diabetes
Brief Title: Closing the Loop in Adults With Type 1 Diabetes - Alcohol Consumption
Acronym: ANGELA02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Dr Mark Evans, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 09/H0306/44
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed loop (algorithm) (Experimental): Subcutaneous delivery of Novorapid insulin, dose calculated by computer-driven control algorithm, based on continuous glucose sensor readings
  Interventions: Device: Closed loop
- Open loop (Placebo Comparator): Subcutaneous delivery of Novorapid insulin according to usual pump regime
  Interventions: Device: Conventional insulin pump delivery

INTERVENTIONS:
Device: Closed loop — Subcutaneous delivery of Novorapid insulin, dose calculated by control algorithm, based on continuous glucose sensor readings
  Arms: Closed loop (algorithm)
Device: Conventional insulin pump delivery — Subcutaneous delivery of Novorapid insulin according to usual pump regime
  Arms: Open loop

SUMMARY:
The main objective is to assess the efficacy and safety of overnight automated closed loop glucose control using a computer-based algorithm compared with conventional insulin pump therapy in adults with type 1 diabetes following the consumption of a moderate amount of alcohol at dinnertime.

DETAILED DESCRIPTION:
People with type 1 diabetes need regular insulin injections or continuous delivery of insulin using an insulin pump. Keeping blood sugars in the normal range is known to reduce the risk of long term complications involving the eyes, kidneys and heart. However, achieving treatment goals can be very difficult as the tighter we try to control blood glucose levels, the greater the risk of the person developing episodes of low glucose levels (hypoglycaemia). One solution is using a system where the amount of insulin injected closely matches the blood sugar levels on a continuous basis. This can be achieved by what is known as a "closed loop system" where a small glucose sensor placed under the skin communicates with a computer containing an algorithm that drives a subcutaneous insulin pump. This system is being developed in Cambridge and is undergoing trials in children and adults with type 1 diabetes. Results thus far show that the system is very effective at preventing hypoglycaemia and maintaining blood glucose levels in target range.

We plan to test the closed loop in various challenging conditions faced by patients in daily life. One of these is the consumption of alcohol, which can give rise to delayed hypoglycaemia in patients with diabetes. The studies will be done in a clinical research facility under supervised conditions. Subjects will attend for two study nights where they will receive a specific volume of alcohol with an evening meal. On one night this will be followed by closed loop algorithm control of their insulin overnight. On the other (control) night subjects will remain on their usual pump therapy regime overnight.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes, as defined by WHO for at least 6 months or confirmed C-peptide negative
* On insulin pump therapy for at least 3 months

Exclusion Criteria:

* Non-type 1 diabetes mellitus
* Any physical/psychological disease likely to interfere with the study
* Taking medication likely to interfere with interpretation of results
* Known/suspected allergy against insulin
* Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator
* Unstable blood glucose control, including recurrent severe hypoglycaemia as judged by the investigator
* Current pregnancy/breastfeeding
* Total daily insulin dose > 1.4 IU/kg
* HbA1C > 10% within the last 3 months
* Unable/unwilling to consume the necessary quantity of alcohol stated in the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Percentage of plasma glucose values in target (3.9-8.0 mmol/L) | 2200-1200hr

SECONDARY OUTCOMES:
Percentage of CGM (continuous glucose monitoring) values in target (3.9-8.0 mmol/L) | 2200-1200; 0000-0400; 0400-0800; 0800-1200; 0300-1200hrs
Percentage of plasma glucose and CGM values in target (3.9-8.0 mmol/L) | 0000-0400; 0400-0800; 0800-1200; 0300-1200hrs
Percentage of plasma glucose and CGM values below 3.9 mmol/L | 2200-1200; 0000-0400; 0400-0800; 0800-1200; 0300-1200hrs
Percentage of plasma glucose and CGM values above 8.0 mmol/L | 2200-1200; 0000-0400; 0400-0800; 0800-1200; 0300-1200hrs
Average plasma and CGM glucose | 2200-1200; 0000-0400; 0400-0800; 0800-1200; 0300-1200hrs
Average plasma insulin concentration | 2200-1200; 0000-0400; 0400-0800; 0800-1200; 0300-1200hrs
Total dose of insulin administered | 2200-1200hrs
Low blood glucose index (LBGI) score | 2200-1200; 0000-0400; 0400-0800; 0800-1200; 0300-1200hrs
High blood glucose index (HBGI) score | 2200-1200; 0000-0400; 0400-0800; 0800-1200; 0300-1200hrs
Percentage of plasma glucose and CGM values below 3.0 mmol/L | 2200-1200; 0000-0400; 0400-0800; 0800-1200; 0300-1200hrs

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Evans, MD FRCP, Principal Investigator — University of Cambridge, UK; Roman Hovorka, PhD, Study Director — University of Cambridge, UK
Locations (1):
- Addenbrooke's Hospital, Cambridge, United Kingdom

REFERENCES:
- [Derived] Hovorka R, Kumareswaran K, Harris J, Allen JM, Elleri D, Xing D, Kollman C, Nodale M, Murphy HR, Dunger DB, Amiel SA, Heller SR, Wilinska ME, Evans ML. Overnight closed loop insulin delivery (artificial pancreas) in adults with type 1 diabetes: crossover randomised controlled studies. BMJ. 2011 Apr 13;342:d1855. doi: 10.1136/bmj.d1855. PMID 21493665